CLINICAL TRIAL: NCT02608970
Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of BMS-986177 in Healthy Subjects
Brief Title: Safety and Tolerability Study of BMS-986177 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV010-001; 2015-003065-29 (EudraCT Number)
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BMS-986177 (Experimental): BMS-986177 specified dose on specified days
  Interventions: Drug: BMS-986177
- Placebo (Other): Placebo specified dose on specified days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986177
  Arms: BMS-986177
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and pharmacokinetics of BMS-986177 in healthy subjects

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs and clinical laboratory determinations
* Body Mass Index (BMI) of 18 to 30 kg/m2 inclusive. BMI = weight (kg)/ [height (m)]2
* Females who are not of childbearing potential (i.e., who are post-menopausal or surgically sterile) and men ages 18 to 55, inclusive

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations beyond what is consistent with the target population
* Any condition that could affect drug absorption
* Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-23 (Actual)

PRIMARY OUTCOMES:
Safety of single dose of BMS-986177 measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Approximately 3 days
  Adverse event (AE), Serious adverse event (SAE)
Safety of multiple dose of BMS-986177 measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Approximately 16 days
Tolerability of single dose of BMS-986177 measured by number of subjects who experience SAEs, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Approximately 3 days
Tolerability of multiple dose of BMS-986177 measured by number of subjects who experience SAE, deaths, AEs leading to discontinuation, and potential clinically significant changes in ECG parameters, vital signs, laboratory tests and physical examinations | Approximately 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- SGS Belgium NV, Antwerp, Belgium

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx